CLINICAL TRIAL: NCT03904394
Title: The Impact of Nitrate-reducing Capacity of Oral Bacteria on Post-exercise Hypotension in Healthy Individuals.
Brief Title: Oral Nitrite Synthesis and Post-exercise Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Raul Bescos, Director, University of Plymouth
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: (16/17)-666
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Blood Pressure; Sports Physical Therapy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Mouthwash (Placebo Comparator)
  Interventions: Other: Exercise
- Antibacterial Mouthwash (Active Comparator)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Four sets of 7 minutes at 65% of VO2peak interspersed with 3 min of passive recovery

SUMMARY:
Exercise is probably the most effective approach to reduce blood pressure. In fact, a single bout of exercise induces a physiological response known as Post-Exercise Hypotension (PEH) where a prolonged decrease in resting blood pressure occurs in the minutes and hours after exercise. However, it is not fully understood how this response triggers. Recent evidence suggests that oral bacteria may play a key role in blood pressure control by enhancing nitrite, and then nitric oxide (NO) bioavailability under resting conditions in humans. However, no previous study has investigated whether this is a key mechanism involve in PEH. Thus, the main aim of this study was to investigate if the oral nitrate/nitrite pathway is a key regulator of PEH and vasodilation in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

Blood pressure (SBP < 130 mmHg; DBP < 90 mmHg) BMI < 30 kg/m2 Age 18 to 50 years old

Exclusion Criteria:

Smoker Hypertension Dyslipidaemia Diabetes Gingivitis or periodontitis Using antibacterial mouthwash or tongue scrapes Taking antibiotics 1 month before the start of the study Females without have irregular menstrual periods

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure after exercise | Baseline and 1 hour and 2 hours after exercise
  Blood pressure was measured before and at 1 hour and 2hours after exercise using an electronic sphygmomanometer (ProBP 3400, Welch Allyn). The second and third readings will be averaged to determine mean blood pressure.

SECONDARY OUTCOMES:
Change in reactive hyperaemia | Baseline and 1 hour and 2 hours after exercise
  Tissue oxygenation index (TOI) were recorded on the left forearm (extensor digitorum) using a NIRS system (NIRO-200NX, Hamamatsu) before exercise and 2 hours after exercise. After baseline measurements (2 minutes), an automatic pneumatic cuff (Hokanson E-20 AG101) was inflated ~5cm above the elbow for 5 minutes to an occlusion pressure of 200 mmHg. Then, inflation of the cuff was rapidly released (< 1 second) and the NIRS measurements were continuously monitored for 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Crai Cutler, MSc, Principal Investigator — University of Plymouth
Locations (1):
- Laboratory of Nutrition, Exercise & Health, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Information will be available upon request